CLINICAL TRIAL: NCT01283178
Title: A Phase I Dose Escalation Trial: Concurrent Intensity-Modulated Radiotherapy (IMRT) and Chemotherapy With Molecular Image-Guided Adaptive Radiation Therapy (IGART) for Advanced Head and Neck Squamous Cell Carcinomas (HNSCC)
Brief Title: Phase I Study of IMRT and Molecular-Image Guided Adaptive Radiation Therapy for Advanced HNSCC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated. The data analysis was futile with only 3 accruals. PI opted to terminate with IRB and withdraw FDA IND.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC 13222; NCI-2010-02340 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016059 (NIH)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Salivary Gland Squamous Cell Carcinoma; Stage II Salivary Gland Cancer; Stage II Squamous Cell Carcinoma of the Hypopharynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Verrucous Carcinoma of the Oral Cavity
Keywords: squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; alovudine; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo intensity-modulated image-guided adaptive radiotherapy once daily 5 days a week for 6 weeks. Patients also receive cisplatin IV on days 1 and 22. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: intensity-modulated radiation therapy; Drug: cisplatin; Radiation: image-guided adaptive radiation therapy; Other: 3'-deoxy-3'-[18F]fluorothymidine; Procedure: positron emission tomography/computed tomography; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Radiation: intensity-modulated radiation therapy — Undergo intensity-modulated image-guided adaptive radiotherapy
  Other Names: IMRT
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Radiation: image-guided adaptive radiation therapy — Undergo intensity-modulated image-guided adaptive radiotherapy
  Other Names: IGART; image-guided adaptive radiotherapy
Other: 3'-deoxy-3'-[18F]fluorothymidine — Undergo FLT-PET scans for IMRT/IGART
  Other Names: 18F-FLT
Procedure: positron emission tomography/computed tomography — Undergo FDG/FLT-PET scans for IMRT/IGARTT
Radiation: fludeoxyglucose F 18 — Undergo FDG-PET scans for IMRT/IGART
  Other Names: 18FDG; FDG

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. CT and PET scans and treatment-planning systems may help in planning radiation therapy. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with cisplatin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of intensity-modulated image guided adaptive radiation therapy when given together with cisplatin in treating patients with locally advanced head and neck squamous cell cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of integrating molecular imaging (PET with FLT tracer) into current state-of-the-art image-guided adaptive radiation therapy (IGART) of head and neck cancer.

II. To determine within a predefined range the maximum tolerated radiation dose for concurrent cisplatin and molecular and anatomic image-based IGART of head and neck cancer.

SECONDARY OBJECTIVES I. To compare gross tumor volumes defined by FDG-PET, FLT-PET, CBCT, and regular FBCT before, during, and following completion of chemo-radiation therapy.

II. To evaluate the impact of escalated doses to tumor sub-volumes with high FLT and FDG uptake prior to and during radiation therapy using post-treatment FDG images as an early surrogate for sub-volume-specific local control.

III. To develop a database consisting of all molecular and anatomic images, including daily CBCT data sets, obtained during chemo-radiation therapy to support further research. Potential applications include determination of optimal adaptive re-planning frequency and the benefits of basing IGART on 4D anatomic data sets derived from deformably registering daily CBCT and FBCT data sets.

IV. Determine patient long-term toxicities and survival. V. To evaluate the impact of daily image-guided setup; off-line every other week adaptive re-planning; and molecular-image based targeting on sparing of tissues and organs responsible for late and early treatment sequelae.

OUTLINE: This a dose-escalation study of intensity-modulated radiotherapy.

Patients undergo intensity-modulated image-guided adaptive radiotherapy once daily 5 days a week for 6 weeks. Patients also receive cisplatin IV on days 1 and 22. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 and 4 weeks, 2, 3, 4, 5, 6, 9, and 12 months, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of head and neck malignancy without clinical or radiographic evidence of metastatic disease
* Locally advanced HN SCC, stages III, IV, and bulky (> 27 cm^3 volume) stage II, excluding larynx and nasopharynx, of no more than 150 cm^3 volume base on CT scan
* All patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines
* Candidate for chemotherapy
* Zubrod performance score of 0 or 1
* Absolute granulocyte count (AGC) >= 2000 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Hemoglobin > 8.0 g/dl based upon CBC/differential obtained within 2 weeks prior to registration on study
* Serum creatinine =< 1.5 mg/dl or measured or calculated creatinine clearance >= 50 ml/min
* Negative pregnancy test within 2 weeks prior to registration for women of childbearing potential

Exclusion Criteria:

* Prior invasive malignancy except non-melanomatous skin cancers unless patient has been disease free for at least 3 years
* Prior cancer treatment for this cancer, including gross total tumor excision
* Prior radiation treatment to the HN region
* Patients with known syndromes that alter radiosensitivity
* Any medical contraindications for chemotherapy
* Pregnant or lactating women
* Women (of childbearing potential) and men who are sexually active and are not willing/able to use a medically acceptable form of contraception throughout the treatment and 60 days thereafter

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of integrating molecular imaging (PET with FLT tracer) into current state-of-the-art image-guided adaptive radiation therapy (IGART) of head and neck cancer | 6 weeks

SECONDARY OUTCOMES:
Comparison of gross tumor volumes defined by FDG-PET, FLT-PET, CBCT, and regular FBCT | Before, during, and following completion of chemoradiation therapy
Impact of escalated doses to tumor sub-volumes with high FLT and FDG uptake using post-treatment FDG images as an early surrogate for sub-volume-specific local control | Prior to and during radiation therapy
Development of a database consisting of all molecular and anatomic images, including daily CBCT data sets, obtained during chemo-radiation therapy to support further research | Up to 5 years
Patient long-term toxicities and survival | At 2 and 4 weeks, 2, 3, 4, 5, 6, 9, and 12 months, every 6 months for 2 years, and then annually for 2 years
Impact of daily image-guided setup; off-line every other week adaptive re-planning; and molecular-image based targeting on sparing of tissues and organs responsible for late and early treatment sequelae | At 2 and 4 weeks, 2, 3, 4, 5, 6, 9, and 12 months, every 6 months for 2 years, and then annually for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shiyu Song, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The data analysis was futile with only 3 accruals. PI opted to terminate with the IRB and withdraw the FDA IND.